CLINICAL TRIAL: NCT00067093
Title: Safety and Efficacy Trial Evaluating the Use of SR34006 in the Treatment of Deep Vein Thrombosis (DVT)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: ICD Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EFC3491; SR34006
Record Dates: First submitted 2003-08-11; First posted 2003-08-13 (Estimated); Last update posted 2011-04-06 (Estimated); Status verified 2011-04

CONDITIONS: Deep Vein Thrombosis
MeSH Terms: conditions — Venous Thrombosis | interventions — idraparinux; Dalteparin; Heparin; acarboxyprothrombin

INTERVENTIONS:
Drug: SanOrg34006
Drug: LMW heparin
Drug: Unfractionated heparin
Drug: Vitamin K antagonist (VKA)

SUMMARY:
Patients who have deep vein thrombosis (blood clot in the leg) will be treated in this study. The purpose of the study is to compare the safety and effectiveness of a new injectable anticoagulant (blood thinning) drug administered once each week, SanOrg34006, with the standard way of treating deep vein thrombosis. The standard treatment includes injections or infusions of an anticoagulant drug (Unfractionated Heparin or low molecular weight heparin) for about a week, followed by vitamin K antagonist (VKA) anticoagulant tablets (warfarin or acenocoumarol) which are taken by mouth. Eligible patients will be assigned to treatment with either SanOrg34006 or the combination of Unfractionated Heparin or low molecular weight heparin plus a VKA (warfarin or acenocoumarol) by random chance. Treatment will be known to both patients and their doctors.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed acute symptomatic DVT
* Written informed consent

Exclusion Criteria:

* Legal lower age limitations
* Patients with symptomatic pulmonary embolism
* Thrombectomy, insertion of a caval filter, or use of a fibrinolytic agent to treat the current episode of DVT
* Other indication for VKA than DVT
* More than 36 hours before the treatment with therapeutic dosages of low molecular weight heparin or initiation of VKA treatment prior to randomization
* Participation in another pharmacotherapeutic study within the prior 30 days
* Creatinine clearance <10mL/min, severe hepatic disease or bacterial endocarditis
* Life expectancy <3 Months
* Active bleeding or high risk for bleeding
* Uncontrolled hypertension: systolic blood pressure >180 mm Hg and diastolic blood pressure >110 mm Hg.
* Pregnancy or childbearing potential without proper contraceptive measures
* Any other contraindication listed in the labeling of warfarin, acenocoumarol, unfractionated heparin (UFH), enoxaparin, or tinzaparin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1452 (Actual)
Dates: Start 2003-05; Primary Completion 2005-09 (Actual); Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
symptomatic recurrent pulmonary embolism or deep vein thrombosis within 3 months

SECONDARY OUTCOMES:
symptomatic recurrent PE/DVT within 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: ICD CSD, Study Director — Sanofi
Locations (24):
- United States (24):
  - University of Colorado Health Sciences Center, Denver, Colorado
  - Jackson Cardio-Vascular Clinic, Jacksonville, Florida
  - MIMA Century Research Associates, Melbourne, Florida
  - Medical College of Georgia, Augusta, Georgia
  - DeKalb Medical Center, Decatur, Georgia
  - Northwestern University, Chicago, Illinois
  - Evanston Northwestern Healthcare, Evanston, Illinois
  - Loyola University of Chicago, Maywood, Illinois
  - Consultants in Pulmonary Medicine, Olathe, Kansas
  - Boston Medical Center, Boston, Massachusetts
  - St. Joseph Mercy - Oakland Research Center, Pontiac, Michigan
  - Lovelace Health Systems, Albuquerque, New Mexico
  - North Shore University Hospital, Manhasset, New York
  - University of Rochester Medical Center, Rochester, New York
  - Health System Research Center, Grand Forks, North Dakota
  - University of Oklahoma HSC, Oklahoma City, Oklahoma
  - Lehigh Valley Hospital, Allentown, Pennsylvania
  - James Muntz, Houston, Texas
  - Scott and White Memorial Hospital & Clinic, Temple, Texas
  - Inova Alexandria Hospital, Alexandria, Virginia
  - Pulmonary Associates, Fredericksburg, Virginia
  - McGuire VAMC, Richmond, Virginia
  - Swedish Medical Center, Seattle, Washington
  - William Dittman, Spokane, Washington

REFERENCES:
- [Derived] Prins MH, Guillemin I, Gilet H, Gabriel S, Essers B, Raskob G, Kahn SR. Scoring and psychometric validation of the Perception of Anticoagulant Treatment Questionnaire (PACT-Q). Health Qual Life Outcomes. 2009 Apr 7;7:30. doi: 10.1186/1477-7525-7-30. PMID 19348685
- [Derived] van Gogh Investigators; Buller HR, Cohen AT, Davidson B, Decousus H, Gallus AS, Gent M, Pillion G, Piovella F, Prins MH, Raskob GE. Idraparinux versus standard therapy for venous thromboembolic disease. N Engl J Med. 2007 Sep 13;357(11):1094-104. doi: 10.1056/NEJMoa064247. PMID 17855670
- See also: Related Info — http://www.sanofi-aventis.com